CLINICAL TRIAL: NCT01292356
Title: Study of Skin Toxicity of Cetuximab: Find a Link Between Skin Inflammation and Tumor Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Docteur David TOUGERON, CHU DE POITIERS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUTACETUX 2010-0198378-85
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

ARMS (1):
- cetuximab (Experimental)
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab

SUMMARY:
Colon cancer is one of the most common cancers in France with more than 36,000 new cases per year. Despite significant advances in therapeutic care, the prognosis of colon cancers with metastases remains bad. The treatment of metastatic disease is based on chemotherapy coupled with therapeutic antibodies. The most commonly used are anti-EGFR (Epidermal Growth Factor Receptor), which allowed a significant increase in patient survival. They are responsible for skin toxicity in the form of an acneiform rash which can be debilitating for patients and require discontinuation of treatment. However, this toxicity is strongly correlated with treatment efficacy. Understanding the mechanisms of cutaneous side effects of anti-EGFR is therefore a major challenge to treat and better understand the association with treatment efficacy.

The objective of this study is to investigate a link between cutaneous inflammatory response in patients treated with anti-EGFR, serum level of anti-EGFR and treatment efficacy. It will be conducted systematic consultations dermatology, skin biopsies and blood samples in patients treated with anti-EGFR. From biopsies, it will be searched by an infiltration of inflammatory cells and expression of genes involved in skin inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patient with histologically proven metastatic colorectal cancer with KRAS wild-type
* Treatment with cetuximab in first line chemotherapy combined with FOLFOX or FOLFIRI
* Patient has signed informed consent
* Patient affiliated to the Social Security
* Prescription of cetuximab in agreement with the Summary of Product Characteristics

Exclusion Criteria:

* Patients aged under 18
* Patients taking immunosuppressive therapy
* Patient having a severe skin disease
* No measurable metastasis
* Patients with a contra-indication of cetuximab: hypersensitivity to cetuximab or to any excipients
* Severe alteration of respiratory or cardiac function or severe coronary disease
* Patients with contra-indication to chemotherapy FOLFOX and FOLFIRI
* Participation in another research protocol
* Patients not affiliated to the Social Security
* Hospitalized patients without consent
* Pregnant or nursing women, women of childbearing age with no effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12-20 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
Main criteria is the variation of skin pro-inflammatory cytokines in pre and post-therapeutic punch skin biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Poitiers, Poitiers, France